CLINICAL TRIAL: NCT03769376
Title: Histologic Comparison of Healing After Tooth Extraction With Ridge Preservation Using Two Different Xenografts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1722
Record Dates: First submitted 2018-11-29; First posted 2018-12-07 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Partial Edentulism
Keywords: toothlessness

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned (1:1) to one of two treatment groups (Bio-Oss® or Salvin-Oss®) at the time of surgery through random selection of sealed envelopes.
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomly assigned (1:1) to one of two treatment groups (Bio-Oss® or Salvin-Oss®) at the time of surgery through random selection of sealed envelopes. The outcome assessor for histological samples will not be aware of which group the participant was in until code unlocked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bio-Oss® (Active Comparator): Bio-Oss® xenograft bone material will be placed into the socket following tooth extraction. Half of participants will be randomly assigned to this treatment group (1:1).
  Interventions: Device: Bio-Oss®
- Salvin-Oss® (Active Comparator): Salvin-Oss® xenograft bone material will be placed into the socket following tooth extraction. Half of participants will be randomly assigned to this treatment group (1:1).
  Interventions: Device: Salvin-Oss®

INTERVENTIONS:
Device: Bio-Oss® — Bio-Oss® xenograft bone material will be placed into the socket following tooth extraction.
  Arms: Bio-Oss®
Device: Salvin-Oss® — Salvin-Oss® xenograft bone material will be placed into the socket following tooth extraction.
  Arms: Salvin-Oss®

SUMMARY:
The purpose of this study is to compare the speed of bone healing of the two most commonly used xenografts on the market, Bio-Oss® and Salvin-Oss® using a tooth extraction ridge preservation model in participants scheduled for tooth extraction and subsequent receipt of a dental implant. Researchers hypothesize that there will be additional vital bone at 16-20 weeks with Salvin-Oss®.

DETAILED DESCRIPTION:
This study focuses on xenografts to preserve alveolar bone after tooth extraction prior to placement of a dental implant. Extraction sites that are not grafted for ridge preservation may lose up to 50 percent of their ridge width the first year after extraction. Xenografts are one of several products on the market used to maintain ridge width after tooth extraction. This study aims to compare the two most commonly used, FDA-approved xenografts on the market, Bio-Oss® and Salvin-Oss, in the preservation of alveolar bone after extraction of non-molar teeth.

The primary objective of this study is to histologically evaluate and compare the percentage of new bone formation in healing extraction sockets of non-molar teeth grafted with Bio-Oss® versus Salvin-Oss®. The secondary aim is to observe clinical changes in ridge height and ridge width after grafting with these two materials.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Consent to be in the study.
* Planned for non-emergent dental treatment.
* American Society of Anesthesiologist Class I or II.
* Require extraction of a single-rooted non-molar tooth.
* Committed to have the dental implant placed at the site of extraction 16-20 weeks after extraction and ridge preservation.
* Adequate restorative space for implant-retained restoration.
* > 10mm alveolar bone height without impingement on the maxillary sinus or inferior alveolar canal.
* Root location and angulation that would be consistent with the subsequent implant placement.
* Roots with minimum of 10mm of radiographic bone support.
* Root angulation similar to the angulation of the implant to be placed at the site.

Exclusion Criteria:

* < 18 years old.
* Currently pregnant.
* Require antibiotic prophylaxis prior to dental procedures as outlined by the 2017 American Heart Association guidelines.
* Decisionally challenged individuals.
* Current smokers.
* American Society of Anesthesiologist Class III or IV.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Font, DDS, MS, Principal Investigator — University of Colorado, Denver; Charles A Powell, DDS, MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado School of Dental Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bio-Oss® | Salvin-Oss®
Started | 20 | 18
Completed | 13 | 11
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: Detailed demographics data was not collected for any participant for this study beyond what was required to be verified to confirm study eligibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bio-Oss® | Salvin-Oss® | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Customized [Count of Participants; unit: Participants] — More specific age demographics information was not collected for any participant.
  Participants
    <18 years | 0 | 0 | 0
    Between 18 and 100 years | 20 | 18 | 38
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/Gender demographics information was not collected for any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: New Bone Formation at Extraction/Xenograft Site Measured by Histological Evaluation at 16-20 Weeks
Description: The amount of new bone formation at the tooth extraction/xenograft site as measured by the percent of vital bone, residual graft, and connective tissue observed in a histological sample (a bone biopsy) obtained at the time of dental implant insertion, 16-20 weeks after extraction.
Time Frame: Baseline to 16-20 weeks
Population: Only participants that completed the study are included in the analysis.
Measure: Mean (Full Range); unit: Percent
Arm/Group | Bio-Oss® | Salvin-Oss®
Number analyzed (Participants) | 13 | 11
Percent
  Vital bone | 29.38 [14.07 to 54.91] | 32.05 [16.53 to 60.63]
  Residual graft | 14.02 [5.32 to 22.30] | 16.56 [5.95 to 50.16]
  Connective Tissue/other | 56.61 [39.74 to 78.51] | 51.39 [20.35 to 69.57]

2. Primary Outcome: New Bone Formation at Extraction/Xenograft Site Measured Clinically With Dental Probe at 16-20 Weeks
Description: The boney ridge height on both the buccal/lingual and width in area of the extraction/xenograft site as measured at time of implant placement with an intra-oral dental probe at 16-20 weeks after extraction. Percent change in ridge width from baseline is reported
Time Frame: Baseline to 16-20 weeks
Population: Only participants that completed the study are included in the analysis.
Measure: Mean (Full Range); unit: Percent
Arm/Group | Bio-Oss® | Salvin-Oss®
Number analyzed (Participants) | 13 | 11
Percent | 15.38 [0 to 100] | 9.09 [0 to 100]

ADVERSE EVENTS:
Time Frame: 20 Weeks
Arm/Group | Bio-Oss® | Salvin-Oss®
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT03769376/Prot_SAP_000.pdf